CLINICAL TRIAL: NCT02252302
Title: The Effects of Inhaled Beta-2-Agonists and Air Pollution on Lung Function and Athletic Capacity
Brief Title: Exercise in Air Pollution and Lung Health in Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Academy of Sport and Exercise Medicine (CASEM) (Unknown); Natural Sciences and Engineering Research Council, Canada (Other); Fraser Basin Council (Unknown)
Responsible Party: Principal Investigator, Michael Koehle, Principal Investigaor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H13-01079
Record Dates: First submitted 2014-09-16; First posted 2014-09-30 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Exercise-induced Bronchoconstriction; Air Pollution
Keywords: Exercise-induced bronchoconstriction; Air pollution; Exercise; Inhaled beta-2-agonist; Cognitive Function
MeSH Terms: conditions — Motor Activity | interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Resting in diesel exhaust following salbutamol inhalation (Active Comparator): Participants will be sitting in an air pollution chamber while being exposed to diesel exhaust (PM2.5 of 300 μg/m3) for a total of 1hour following the inhalation of 400ug of salbutamol.
  Interventions: Other: Rest (Sitting on chair); Drug: Salbutamol inhalation; Other: Diesel Exhaust Exposure
- Resting in diesel exhaust following placebo inhalation (Placebo Comparator): Participants will be sitting in an air pollution chamber while being exposed to diesel exhaust (PM2.5 of 300 μg/m3) for a total of 1hour following the inhalation of a placebo.
  Interventions: Other: Rest (Sitting on chair); Drug: Placebo inhalation; Other: Diesel Exhaust Exposure
- Cycling in diesel exhaust following salbutamol inhalation (Active Comparator): Participants will be cycling while being exposed to diesel exhaust (PM2.5 of 300 μg/m3) for a total of 1 hr following the inhalation of 400ug of salbutamol.
  Interventions: Other: Cycling exercise; Drug: Salbutamol inhalation; Other: Diesel Exhaust Exposure
- Cycling in diesel exhaust following placebo inhalation (Placebo Comparator): Participants will be cycling while being exposed to diesel exhaust (PM2.5 of 300 μg/m3) for a total of 1 hr following the inhalation of a placebo
  Interventions: Other: Cycling exercise; Drug: Placebo inhalation; Other: Diesel Exhaust Exposure
- Resting in filtered air following salbutamol inhalation (Sham Comparator): Participants will be sitting while being exposed to filtered air for a total of 1hour following the inhalation of 400ug of salbutamol.
  Interventions: Other: Rest (Sitting on chair); Other: Filtered air
- Resting in filtered air following placebo inhalation (Placebo Comparator): Participants will be sitting while being exposed to filtered air for a total of 1hour following the inhalation of a placebo.
  Interventions: Other: Rest (Sitting on chair); Other: Filtered air
- Cycling in filtered air following salbutamol inhalation (Sham Comparator): Participants will be cycling while being exposed to filtered air for a total of 1 hr following the inhalation of 400ug of salbutamol.
  Interventions: Other: Cycling exercise; Drug: Salbutamol inhalation; Other: Filtered air
- Cycling in filtered air following placebo inhalation (Placebo Comparator): Participants will be cycling while being exposed to filtered air for a total of 1 hr following the inhalation of a placebo
  Interventions: Other: Cycling exercise; Drug: Placebo inhalation; Other: Filtered air

INTERVENTIONS:
Other: Rest (Sitting on chair) — Study participants will sit on a chair for 60min. This is to simulate physical resting condition.
  Arms: Resting in diesel exhaust following placebo inhalation; Resting in diesel exhaust following salbutamol inhalation; Resting in filtered air following placebo inhalation; Resting in filtered air following salbutamol inhalation
Other: Cycling exercise — Study participants will exercise on a cycle ergometer for 45min. Participants will start their 30-min long constant workload exercise test test 60-min after the drug intervention. The exercise test will be set to a resistance of 50% of the maximal wattage that was reached on the graded exercise test on the screening day. The cycling exercise intervention will follow the rest-intervention.
  Arms: Cycling in diesel exhaust following placebo inhalation; Cycling in diesel exhaust following salbutamol inhalation; Cycling in filtered air following placebo inhalation; Cycling in filtered air following salbutamol inhalation
Drug: Salbutamol inhalation — Study participants will be exposed to 400ug of salbutamol prior to entering the air pollution chamber.
  Arms: Cycling in diesel exhaust following salbutamol inhalation; Cycling in filtered air following salbutamol inhalation; Resting in diesel exhaust following salbutamol inhalation
Drug: Placebo inhalation — Study participants will inhale a placebo (placebo for salbutamol) prior to entering the air pollution chamber
  Arms: Cycling in diesel exhaust following placebo inhalation; Cycling in filtered air following placebo inhalation; Resting in diesel exhaust following placebo inhalation
Other: Diesel Exhaust Exposure — Participants will be exposed to PM2.5 of 300 μg/m3
  Arms: Cycling in diesel exhaust following placebo inhalation; Cycling in diesel exhaust following salbutamol inhalation; Resting in diesel exhaust following placebo inhalation; Resting in diesel exhaust following salbutamol inhalation
Other: Filtered air — Participants will be breathing filtered air
  Arms: Cycling in filtered air following placebo inhalation; Cycling in filtered air following salbutamol inhalation; Resting in filtered air following placebo inhalation; Resting in filtered air following salbutamol inhalation

SUMMARY:
When exposed to air pollution, the asthma symptoms are aggravated and lung function is impaired. Due to high breathing rates and volumes, physically active individuals are at particular risk of lung health impairment due to the high breathing rates and volumes. Greater doses of air pollutants reach deeper areas in the lungs where they can trigger asthma-symptoms. When treating these symptoms with inhaled beta-2-agonists the airways widen even more, allowing the air pollutants to reach even deeper areas of the lung. With this study the investigators investigate how inhaled beta-2-agonists affect athletic capacity and lung health in physically active asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* mild-moderate asthmatics with controlled treatment (definition of "mild": percent fall index at eucapnic voluntary hyperpnea (EVH) test on screening day between 10-15%; "moderate": percent fall index at EVH test on screening day between 15 - 20%).
* men and non-pregnant women

Exclusion Criteria:

* any history of uncontrolled respiratory or cardiac disease
* pregnancy
* allergic reactions to lidocaine and salbutamol
* any recent infections or orthopaedic nasal issues/injuries that may interfere with the insertion of the catheter needed to assess expiratory flow limitation or work of breathing
* claustrophobia in small rooms, comparable to the air pollution chamber used for this study.
* English as a second language (ESL) - participants who are not able to understand the risk that may be associated with the participation in this study due to language difficulties after following the University of British Clinical Research Ethics Board Guidance Notes 13.2.1. (ESL participants will be given a consent form in the most appropriate language or an appropriate translator will be present during the initial consent process).

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in rating of perceived exertion for breathing, dyspnea | Difference in perceived dyspnea between salbutamol and placebo exposure as well as polluted air and filtered air. Dyspnea ratings will be collected every 2.5min for a duration of 45min during the exercise test.

SECONDARY OUTCOMES:
Change in work of breathing (WOB) between filtered air and polluted air | work of breathing will be assessed every 2.5min for a time period of 45min during the exercise bout

OTHER OUTCOMES:
Change in spirometry (FEV1 and FVC) between filtered air and polluted air | Spirometry will be assessed at baseline and 45min after the start of the exercise bout.
Change in cognitive function | Cognitive function will be assessed at baseline (prior to entering the air pollution chamber) and 45 min after the start of the exercise intervention.
  cognitive function will be assessed using the NIH toolbox tests and the brain derived neurotrophic factor (BDNF) blood serum measurements
Retinal Imaging | The retina will be imaged at baseline (prior to entering the air pollution chamber) and 20 min after the completion of the exercise intervention.
  The blood vessels in the eye will be imaged using a camera.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Koehle, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Environmental Physiology Laboratory, Vancouver, British Columbia, Canada